CLINICAL TRIAL: NCT06705946
Title: Effects of Dynamic Stability Training Using Water Inertia Load on Lower Limb Joint Moments, Gait and Balance in Elderly Women
Brief Title: Effects of Water Inertia Load Training on Lower Limb Joint Moments, Gait, and Balance in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hyun Ju Kim (Other)
Responsible Party: Sponsor-Investigator, Hyun Ju Kim, Principal Investigator, Busan University of Foreign Studies
Organization: Busan University of Foreign Studies (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUFS-DST-2024
Record Dates: First submitted 2024-11-23; First posted 2024-11-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Balance and Gait Impairment in Elderly Women
Keywords: elderly women; gait; balance; dynamic stability training; water Inertia Load

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aqua vest group (Experimental): Participants in this group will perform Dynamic Stability Training (DST) sessions twice a week for 12 weeks while wearing an aqua vest. Each session will focus on dynamic stability exercises aimed at improving balance, lower limb joint moment distribution, and gait. Each session will last for 50 minutes
  Interventions: Behavioral: Aqua vest group
- Weight vest group (Active Comparator): Participants in this group will perform the same Dynamic Stability Training (DST) sessions twice a week for 12 weeks, but with a weight vest instead of an aqua vest. Each session will focus on balance, lower limb joint moment distribution, and gait, lasting for 50 minutes
  Interventions: Behavioral: Weight vest group

INTERVENTIONS:
Behavioral: Aqua vest group — Participants in this group will perform Dynamic Stability Training (DST) sessions twice a week for 12 weeks while wearing an aqua vest. Each session will focus on dynamic stability exercises aimed at improving balance, lower limb joint moment distribution, and gait. Each session will last for 50 minutes
  Arms: Aqua vest group
Behavioral: Weight vest group — Participants in this group will perform the same Dynamic Stability Training (DST) sessions twice a week for 12 weeks, but with a weight vest instead of an aqua vest. Each session will focus on balance, lower limb joint moment distribution, and gait, lasting for 50 minutes
  Arms: Weight vest group

SUMMARY:
This study highlights that age-related neuromuscular changes negatively impact muscle strength, balance, joint mobility, and cardiovascular health, which in turn affect daily life activities and independence. In particular, aging leads to slower gait speeds and increased metabolic costs associated with shifting the body's center of mass, which are closely linked to functional decline in older adults. While previous studies have focused primarily on spatiotemporal variables like stride length and walking speed, there is a lack of research examining exercise interventions that analyze lower limb joint moments. This study aims to assess the effects of dynamic stability training using water inertia load on the distribution of lower limb joint moments, gait, and balance in older adults, ultimately providing valuable insights to support improvements in efficient gait function among the elderly.

DETAILED DESCRIPTION:
1. Study Participants

   This study targets healthy women aged 65 and older who have not engaged in regular exercise in the past six months. Participants will be recruited through posted announcements at Mirine Center and Busan University of Foreign Studies in Busan. Individuals who express interest and sign the consent form after being informed of the study's purpose and eligibility criteria will be selected as participants.

   The appropriate sample size was determined using G*Power 3.1 software, with an effect size of 0.32, a power of 0.8, and a significance level of 0.05, resulting in an estimated sample size of 18 participants. However, to account for potential dropouts, the study will proceed with a total of 30 participants, divided into 15 in the experimental group and 15 in the control group. Participants will be randomly assigned to either the experimental or control group on the first day of exercise at a 1:1 ratio.
2. Measurement

   1. Balance Measurement For this study, a ground reaction force plate (AMTI-OR6, Watertown, MA, USA) will be used to evaluate static balance. The device assesses the range, velocity, and Root Mean Square (RMS) of the center of pressure (COP) using pressure sensors.

      To prevent visual distractions during balance assessment, the surrounding environment will be blocked off with curtains. Both legs will be evaluated. For the single-leg standing test, participants will be instructed to stand barefoot, with arms crossed in front of their chest, supporting one leg while lifting the other leg with the knee bent at a 90-degree angle, maintaining the position for 40 seconds.

      This duration was set at 40 seconds to ensure sufficient time for data collection and to remove any errors at the beginning and end of the trial. To ensure accurate results, participants will be given sufficient rest between attempts, and the test will only be conducted once the participant feels fully prepared. Given that it may be challenging for elderly individuals to maintain this position for the full duration, if they cannot reach 40 seconds, the longest time achieved out of five attempts will be averaged for analysis.
   2. Gait Measurement

      In this study, gait spatial and temporal assessments will be conducted using a 6-meter walkway and six 3D infrared motion capture cameras (Vicon camera MX-T20, Oxford Metrics, Oxford, UK).

      The measured variables include cadence, step time, stride time, walking speed, step length, stride length, foot-off timing, single support time, and double support time. Gait measurements will be conducted in an environment free of external distractions.

      Participants will perform several practice walks at their preferred walking speed until they become accustomed to the evaluation. Once a normal walking speed is achieved, three trials will be recorded. Additionally, sufficient rest will be provided between each trial to ensure accurate data collection.
   3. kinetic Measurement

   To evaluate lower limb joint moments, this study will use a 6-meter walkway, six 3D infrared motion capture cameras (Vicon camera MX-T20, Oxford Metrics, Oxford, UK), and sixteen reflective markers (14mm). The reflective markers will be attached to the following anatomical landmarks: bilateral anterior superior iliac spines, posterior superior iliac spines, mid-thigh lateral sides, lateral femoral epicondyles, mid-shanks, lateral malleoli, second metatarsals, and heels. For analysis, participants' height, weight, leg length, and knee and ankle joint widths will be measured and input into the system.

   The analysis will track the movement of reflective markers to calculate hip and ankle joint moments and angular velocities using the Vicon Plug-in Gait system at a sampling rate of 100Hz. Hip and ankle joint moments will be analyzed for maximum moment, average values, and positive work during the terminal stance phase of the gait cycle. Each joint moment will be categorized into flexion and extension moments for analysis.
3. Dynamic Stability Training

   The Dynamic Stability Training (DST) program is based on the Instability Neuromuscular Training program proposed by Kang (2024) and consists of exercises structured in progressive stages. The program spans 12 weeks, with two sessions per week, totaling 24 sessions. Each session lasts 50 minutes and includes a 10-minute warm-up, 30 minutes of DST exercises, and a 10-minute cool-down.

   From weeks 0 to 6, the DST program focuses on bilateral support and weight shifting. From weeks 7 to 12, the exercises progress to include single-leg support movements to enhance balance on one leg, while also increasing speed to adjust exercise intensity. The program incorporates movements involving a step box.

   Each exercise adheres to the ACSM exercise guidelines. During weeks 0 to 6, exercises are performed at low intensity (RPE 9-11) for 30 seconds of activity with 60 seconds of rest, totaling two sets using a weight of 3 kg. From weeks 7 to 12, exercises are conducted at moderate intensity (RPE 12-13) for 45 seconds of activity with 90 seconds of rest, totaling one set using a weight of 4 kg. Rest time between sets is 1 minute.

   The experimental group wears an aqua vest filled with water, while the control group wears a weight vest, performing the same exercises. The load of water and weights is determined based on the Rating of Perceived Exertion (RPE).

   The training sessions will be led by the researcher of this study, who has 13 years of experience. Additionally, two assistant instructors will be assigned to monitor participants throughout the sessions, as the participants are elderly individuals.
4. Statistical Analysis

All data collected in this study will be analyzed using SPSS 28.0 to calculate means and standard deviations. The Shapiro-Wilks test will assess the normality of participants' general characteristics and variables. An independent t-test will verify group homogeneity. To compare intervention effects between groups and changes before, during, and after the intervention within groups, a two-way repeated measures ANOVA will be applied. All statistical significance levels will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women over the age of 65

Exclusion Criteria:

* Musculoskeletal injury within the last 3 months Severe cardiopulmonary disease (heart failure, myocardial infarction) Use of anxiolytics, antidepressants, or sedatives Chronic lung disease Surgery within the last 6 months

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Change in step | 6 weeks and 12 weeks after baseline
  Step time is measured in seconds using a 3D motion capture system
Change in stride time | 6 weeks and 12 weeks after baseline
  Stride time is measured in seconds using a 3D motion capture system.
Change in walking speed | 6 weeks and 12 weeks after baseline
  Walking speed is measured in meters per second using a 3D motion capture system.
Change in cadence | 6 weeks and 12 weeks after baseline
  Cadence is measured in steps per minute using a 3D motion capture system
Change in foot off | 6 weeks and 12 weeks after baseline
  Foot off is measured as a percentage of the gate cycle using a 3D motion capture system.
Change in step length | 6 weeks and 12 weeks after baseline
  Step length is measured in meters per second (m/s) using a 3D motion capture system
Change in stride length | 6 weeks and 12 weeks after baseline
  Stride length is measured in meters per second (m/s) using a 3D motion capture system
Change in single support phase | 6 weeks and 12 weeks after baseline
  The single support phase of the gait cycle is measured as a percentage using a 3D motion capture system
Change in dubble support phase | 6 weeks and 12 weeks after baseline
  The double support phase of the gait cycle is measured as a percentage using a 3D motion capture system
Change in balance stability | 6 weeks and 12 weeks after baseline
  Balance was assessed using a single-leg stance test, measuring the center of pressure(COP) sway in both anterior posterior (AP) and medial-lateral (ML) directions.
Change in Lower limb joint moments | 6 weeks and 12 weeks after baseline
  The moments of the lower limb joints, specifically at the hip and ankle, are measured

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Ju Kim, MSc, Principal Investigator — Department of Sports and Health Convergence
Locations (1):
- University of Foreign Studies of Busan, Busan, Geumjeong-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared via Figshare. The data will include demographic information, raw data from the assessments, and any other relevant data collected during the study.
Supporting Information: SAP
Time Frame: The data will be available immediately after the publication of the study results and will be accessible for at least 5 years
Access Criteria: The data will be openly available via Figshare without the need for a data access request

REFERENCES:
- [Background] Laughton CA, Slavin M, Katdare K, Nolan L, Bean JF, Kerrigan DC, Phillips E, Lipsitz LA, Collins JJ. Aging, muscle activity, and balance control: physiologic changes associated with balance impairment. Gait Posture. 2003 Oct;18(2):101-8. doi: 10.1016/s0966-6362(02)00200-x. PMID 14654213
- [Background] Karamanidis K, Arampatzis A. Mechanical and morphological properties of different muscle-tendon units in the lower extremity and running mechanics: effect of aging and physical activity. J Exp Biol. 2005 Oct;208(Pt 20):3907-23. doi: 10.1242/jeb.01830. PMID 16215218
- [Background] Narici MV, Maffulli N, Maganaris CN. Ageing of human muscles and tendons. Disabil Rehabil. 2008;30(20-22):1548-54. doi: 10.1080/09638280701831058. PMID 18608375
- [Background] Kang HG, Dingwell JB. Dynamics and stability of muscle activations during walking in healthy young and older adults. J Biomech. 2009 Oct 16;42(14):2231-7. doi: 10.1016/j.jbiomech.2009.06.038. Epub 2009 Aug 6. PMID 19664776
- [Background] Chale-Rush A, Guralnik JM, Walkup MP, Miller ME, Rejeski WJ, Katula JA, King AC, Glynn NW, Manini TM, Blair SN, Fielding RA. Relationship between physical functioning and physical activity in the lifestyle interventions and independence for elders pilot. J Am Geriatr Soc. 2010 Oct;58(10):1918-24. doi: 10.1111/j.1532-5415.2010.03008.x. Epub 2010 Aug 24. PMID 20738437
- [Background] Rygiel KA, Picard M, Turnbull DM. The ageing neuromuscular system and sarcopenia: a mitochondrial perspective. J Physiol. 2016 Aug 15;594(16):4499-512. doi: 10.1113/JP271212. Epub 2016 May 7. PMID 26921061
- [Background] Mayfield DL, Cronin NJ, Lichtwark GA. Understanding altered contractile properties in advanced age: insights from a systematic muscle modelling approach. Biomech Model Mechanobiol. 2023 Feb;22(1):309-337. doi: 10.1007/s10237-022-01651-9. Epub 2022 Nov 6. PMID 36335506
- [Background] Newman AB, Visser M, Kritchevsky SB, Simonsick E, Cawthon PM, Harris TB. The Health, Aging, and Body Composition (Health ABC) Study-Ground-Breaking Science for 25 Years and Counting. J Gerontol A Biol Sci Med Sci. 2023 Oct 28;78(11):2024-2034. doi: 10.1093/gerona/glad167. PMID 37431156
- [Background] Cooper R, Kuh D, Cooper C, Gale CR, Lawlor DA, Matthews F, Hardy R; FALCon and HALCyon Study Teams. Objective measures of physical capability and subsequent health: a systematic review. Age Ageing. 2011 Jan;40(1):14-23. doi: 10.1093/ageing/afq117. Epub 2010 Sep 15. PMID 20843964
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966